CLINICAL TRIAL: NCT02535169
Title: Lifestyle-Related Health Outcomes in Prediabetes and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Nana Gletsu Miller, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1403986016
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Prediabetic State; Type 2 Diabetes
Keywords: at risk for type 2 diabetes; currently has type 2 diabetes
MeSH Terms: conditions — Obesity; Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Education and Coaching (Experimental): 1. To evaluate whether a health education and coaching strategy in overweight and obese adolescents (≥85th percentile) with high risk for type 2 diabetes is superior to usual care (single nutrition consultation) for weight management, clinical health outcomes (measures of glucose tolerance), lifestyle behavior outcomes (diet and physical activity) and outcomes of importance to patients such as satisfaction with the health care team, treatment goals, and psychosocial functioning.
  Interventions: Behavioral: Health Education and Coaching Strategy
- Usual Care (Placebo Comparator): 1. Dietary consult only
  Interventions: Behavioral: Dietary consult

INTERVENTIONS:
Behavioral: Health Education and Coaching Strategy — Utilizing health education and health coaching to intervene with adolescents who are at high risk for type 2 diabetes or prediabetes regarding nutrition and physical activity. A 16-week curriculum will be utilized and phone-based coaching visits will be performed.
  Arms: Health Education and Coaching
Behavioral: Dietary consult — A routine clinic-based dietary consult will be performed (approximately 1-hour).
  Arms: Usual Care

SUMMARY:
This study looks as how a health education intervention strategy effects health outcomes in overweight and obese adolescents.

DETAILED DESCRIPTION:
This study aims to do the following:

1. To evaluate whether a health education and coaching strategy in overweight and obese adolescents (≥85th percentile) with high risk for type 2 diabetes is superior to usual care (single nutrition consultation) for weight management, clinical health outcomes (measures of glucose tolerance), lifestyle behavior outcomes (diet and physical activity) and outcomes of importance to patients such as satisfaction with the health care team, treatment goals, and psychosocial functioning.
2. To evaluate whether a health education and coaching strategy in obese adolescents with diabetes (type 1 or type 2) is superior to usual care (single nutrition consultation) for weight management, clinical health outcomes (measures of diabetes control), lifestyle behavior outcomes (diet and physical activity) and outcomes of importance to patients such as satisfaction with the health care team, treatment goals, and psychosocial functioning.
3. At baseline, before the interventions described in Aims 1 and 2, to identify key diet and physical activity factors, patient characteristics, or biomarkers which are predictive of diabetes risk.
4. At baseline, before the interventions described in Aims 1 and 2, can associations between glycemia, cardiometabolic risk factors, and diet and physical activity behaviors in overweight and obese adolescents who are at risk for type 2 diabetes be identified using the Bright Futures questionnaire, a survey for lifestyle behavior which is normally used in the clinic setting.

ELIGIBILITY:
Inclusion Criteria:

1. male and female adolescents/young adults,
2. age 10-21,
3. Tanner stage II-V,
4. overweight or obese (body mass index ≥85th percentile for age and sex).

Exclusion Criteria:

1. pregnancy,
2. use of medications that adversely affect glucose metabolism (such as glucocorticoid-containing medications or atypical antipsychotics), and
3. syndromic obesity (such as Prader Willi, hypothalamic obesity, or Laurence- Moon-Biedl).

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2014-05; Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in the oral disposition index measured by oral glucose tolerance test | 6 months
  oral disposition index = insulinogenic index x 1/fasting insulin

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Hannon, MD, MS, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via presentations and publications.

REFERENCES:
- [Derived] Wagner KA, Armah SM, Smith LG, Pike J, Tu W, Campbell WW, Boushey CJ, Hannon TS, Gletsu-Miller N. Associations between Diet Behaviors and Measures of Glycemia, in Clinical Setting, in Obese Adolescents. Child Obes. 2016 Oct;12(5):341-7. doi: 10.1089/chi.2015.0232. Epub 2016 May 2. PMID 27135792